CLINICAL TRIAL: NCT04658199
Title: An Open-Label Extension Study to Evaluate the Safety and Tolerability of Long-Term UCB0107 Administration in Study Participants With Progressive Supranuclear Palsy
Brief Title: A Study to Test the Safety and Tolerability of Long-term UCB0107 Administration in Study Participants With Progressive Supranuclear Palsy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSP002; U1111-1304-3004 (Other: Universal Trial Number (UTN)); 2024-510951-36 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive supranuclear palsy; UCB0107; Phase 1B study; PSP; Bepranemab
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCB0107 (bepranemab) (Experimental): Subjects in this study arm will receive Intravenous UCB0107.
  Interventions: Drug: UCB0107 (bepranemab)

INTERVENTIONS:
Drug: UCB0107 (bepranemab) — UCB0107 (bepranemab) will be administered in a predefined dosage. Pharmaceutical Form: Solution for infusion Route of Administration: Intravenous

SUMMARY:
The purpose of the study is to assess the long-term safety and tolerability of UCB0107 in study participants with progressive supranuclear palsy (PSP).

ELIGIBILITY:
Inclusion Criteria:

* Participant meets the criteria for possible or probable progressive supranuclear palsy (PSP) Richardson's Syndrome according to the Movement Disorder Society-PSP criteria (Hoeglinger et al, 2017)
* Participant completed the Treatment Period (regardless of the total number of infusions) in PSP003 (NCT04185415)
* Participant can be male or female

  a) A male participant must agree to use contraception as detailed in the protocol during the Treatment Period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period b) A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: I. Not a woman of childbearing potential (WOCBP) OR II. A WOCBP who agrees to follow the contraceptive guidance in the protocol during the Treatment Period and for at least 6 months after the last dose of study treatment.
* Participant (or legal representative, as applicable and acceptable by local regulations) is giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol. Informed consent must be obtained before initiating any study procedures

Exclusion Criteria:

* Participant has met a mandatory withdrawal and/or stopping criterion in PSP003 (NCT04185415)
* Participant made a suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt) during PSP003 (NCT04185415), or has current suicidal ideation with at least some intent to act as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Since Last Visit" version of the Columbia Suicide Severity Rating Scale (CSSRS) at the Day 1 Visit. However, participants will not be excluded if, based upon a mental healthcare professional assessment, and the investigator's judgment of benefit/risk, the participant is deemed suitable for receiving study medication

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2027-12-13 (Estimated); Study Completion 2027-12-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events from Baseline of the open-label extension to the end of the study | From Baseline of the open-label extension to end of study visit (up to 7 years)
  An adverse event (AE) is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory finding) in study participants, users, or other persons, whether or not related to the investigational medicinal product (IMP).

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (11):
- Belgium (2):
  - Psp002 40122, Edegem
  - Psp002 40002, Leuven
- Germany (4):
  - Psp002 40277, Bochum
  - Psp002 40276, Düsseldorf
  - Psp002 40278, Essen
  - Psp002 40024, Hanover
- Spain (3):
  - Psp002 40267, Barcelona
  - Psp002 40100, Madrid
  - Psp002 40268, Pamplona
- United Kingdom (2):
  - Psp002 40175, London
  - Psp002 40165, Southampton

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.